CLINICAL TRIAL: NCT00650936
Title: Closure of Atrial Septal Defects With the AMPLATZER Septal Occluder - Post Approval Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGA-014
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Atrial Septal Defect
Keywords: Atrial; Septal; Defect
MeSH Terms: conditions — Heart Septal Defects, Atrial | interventions — Septal Occluder Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMPLATZER Septal Occluder (Other): Subjects were enrolled if the implant of the AMPLATZER Septal Occluder device was completed or was attempted (delivery system entered the subject's body).
  Interventions: Device: AMPLATZER Septal Occluder

INTERVENTIONS:
Device: AMPLATZER Septal Occluder — AMPLATZER Septal Occluder

SUMMARY:
The purpose of this study is to prospectively evaluate the incidence of hemodynamic compromise and to obtain long-term survival data on patients with the AMPLATZER Septal Occluder

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all inclusion criteria. A patient meets inclusion criteria if he/she:

  * is indicated for implantation with the AMPLATZER Septal Occluder for occlusion of a secundum atrial septal defect (Note: This does not include the indication for closure of a fenestration following a fenestrated Fontan procedure),
  * is willing and able to complete the follow-up requirements of this study, and
  * signs the informed consent (or a legal representative signs the informed consent).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2007-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (51):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Permanente, Los Angeles, California
  - Children's Hospital of Central California, Madera, California
  - Children's Hospital Oakland, Oakland, California
  - University of California, San Francisco, San Francisco, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Jacksonville Pediatric Cardiovascular Center, Jacksonville, Florida
  - Miami Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Hope Children's Hospital, Oak Lawn, Illinois
  - Indiana University, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kentucky, Lexington, Kentucky
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Washington University, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Schneider Children's Hospital, New Hyde Park, New York
  - The New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Children's Hospital of New York-Presbyterian, New York, New York
  - Children's Hospital at Strong, Rochester, New York
  - Sanger Heart & Vascular Institute/Carolinas Medical Center, Charlotte, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - The Children's Hospital at Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital, Oklahoma City, Oklahoma
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Moffitt Heart and Vascular Group, Wormleysburg, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University-Children's, Nashville, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - North Austin Medical Center, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Universtiy of Virginia, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Sacred Heart Children's Hospital, Spokane, Washington
  - Aurora Health Care, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Turner DR, Owada CY, Sang CJ Jr, Khan M, Lim DS. Closure of Secundum Atrial Septal Defects With the AMPLATZER Septal Occluder: A Prospective, Multicenter, Post-Approval Study. Circ Cardiovasc Interv. 2017 Aug;10(8):e004212. doi: 10.1161/CIRCINTERVENTIONS.116.004212. PMID 28801537

RESULTS

PARTICIPANT FLOW:
Groups:
- AMPLATZER Septal Occluder: The single-arm subjects were enrolled if the implant of the AMPLATZER Septal Occluder device was completed or was attempted (delivery system entered the subject's body).
Period: Overall Study
Arm/Group | AMPLATZER Septal Occluder
Started | 1000
Completed | 930
Not Completed | 70

BASELINE CHARACTERISTICS:
Arm/Group | AMPLATZER Septal Occluder
Number analyzed (Participants) | 1000
Age, Continuous [Mean (Full Range); unit: years] | 21 [0.3 to 83.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 649
  Male | 351
Height [Mean (Full Range); unit: centimeters] | 135.3 [33.3 to 198.1]
Weight [Mean (Full Range); unit: kilograms] | 45 [4.5 to 179.2]
Qp/Qs [Mean (Full Range); unit: ratio] — The magnitude of a cardiac shunt is described using Qp/Qs (pulmonary flow/systemic flow).
  ratio | 2.1 [0.0 to 8.3]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Subjects With Two-year Device-related Hemodynamic Compromise
Description: The primary efficacy endpoint was the two-year incidence rate of device-related hemodynamic compromise.
Time Frame: 24 months
Population: The analysis population for the primary efficacy endpoint was all subjects who either reached their two-year visit or had a device-related hemodynamic compromise event.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMPLATZER Septal Occluder
Number analyzed (Participants) | 928
percentage of participants | 0.65 [NA to 1.4] — One-sided analysis conducted and reported in the final report

2. Primary Outcome: Co-Primary Effectiveness Endpoint
Description: The percentage of subjects for whom closure success is achieved through two-years. To meet this endpoint, two criteria must be met:
  Technical Success: Successful deployment of the device percutaneously Closure Success: Closure of the atrial septal defect (i.e., a shunt < 2mm) without the need for surgical repair
Time Frame: 24 months
Population: The analysis population for the co-primary effectiveness endpoint was all subjects who either reached their two-year visit or demonstrated closure of the atrial septal defect prior to or at their 2-year visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMPLATZER Septal Occluder
Number analyzed (Participants) | 987
percentage of participants | 97.87 [96.8 to 98.7]

3. Primary Outcome: Co-Primary Safety Endpoint
Description: The co-primary safety endpoint was the percentage of subjects experiencing a device or delivery system related adverse event
Time Frame: 24 months
Population: The analysis population for the co-primary safety endpoint is all subjects who either reached their two-year visit or had a device or delivery system related adverse event prior to their 2-year visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AMPLATZER Septal Occluder
Number analyzed (Participants) | 930
percentage of participants | 6.34 [4.86 to 8.11]

ADVERSE EVENTS:
Arm/Group | AMPLATZER Septal Occluder
Serious Adverse Events (participants affected / at risk) | 57/1000
Other Adverse Events (participants affected / at risk) | 489/1000
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMPLATZER Septal Occluder (N=1000)
Abnormal Lab Value (General disorders) | 1 (1)
Acute Life Threatening Event (General disorders) | 1 (1)
Acute Subdural Hematoma (General disorders) | 1 (1)
Air Embolus (General disorders) | 1 (1)
Anemias (General disorders) | 1 (1)
Aortic Aneurysms (General disorders) | 1 (1)
Arteriovenous (AV) Fistula (General disorders) | 1 (1)
Aspiration Pneumonia/Necrotizing Pneumonia/Aspiration of Vomitus (General disorders) | 1 (1)
Atrial Ectopic Beats/Premature Atrial Beats/Premature Atrial Contractions/Ectopic Atrial Rhythm (General disorders) | 1 (1)
Atrial Fibrillation (General disorders) | 6 (6)
Atrial Flutter (General disorders) | 3 (3)
Bleeding (General disorders) | 2 (2)
Breath Holding Spell (General disorders) | 1 (1)
Cancer (General disorders) | 1 (1)
Cardiac Arrest (General disorders) | 2 (2)
Cardiac Erosion (General disorders) | 2 (2)
Chest Pain (General disorders) | 2 (2)
Chronic Obstructive Pulmonary Disease (COPD) (General disorders) | 1 (1)
Congestive Heart Failure (General disorders) | 3 (3)
Device Embolization (General disorders) | 4 (4)
Diabetes Mellitus (General disorders) | 1 (1)
Elective Procedure (General disorders) | 2 (2)
Elective Surgery (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
First Degree Heart/AV Block/Cardiac Arrhythmia - 1st degree AV Block (General disorders) | 1 (1)
Gastroenteritis (General disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Hematuria (General disorders) | 1 (1)
Hypotension (General disorders) | 2 (2)
Hypoxemia (General disorders) | 1 (1)
Migraine (General disorders) | 2 (2)
Numbness (General disorders) | 1 (1)
Palpitations (General disorders) | 1 (1)
Pericardial Effusion (General disorders) | 4 (4)
Pericarditis (General disorders) | 1 (1)
Pleural Effusion (General disorders) | 1 (1)
Pneumonia (General disorders) | 1 (1)
Presyncope (General disorders) | 1 (1)
ST Segment Changes (General disorders) | 1 (1)
SVC Syndrome (General disorders) | 1 (1)
Sepsis (General disorders) | 1 (1)
Sinus Bradycardia/Sinus Bradycardia (Cardiac Arrhythmia) (General disorders) | 1 (1)
Stridor (General disorders) | 1 (1)
Stroke (General disorders) | 1 (1)
Surgical Closure of ASD (General disorders) | 7 (7)
Syncope (General disorders) | 1 (1)
Tingling (General disorders) | 1 (1)
VASC Pseudoaneurysm (General disorders) | 1 (1)
Vaso Vagal Response (General disorders) | 1 (1)
Visual Disturbance (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMPLATZER Septal Occluder (N=1000)
AV Block (Cardiac disorders) | 1 (1)
Abdominal Pain (General disorders) | 10 (11)
Abdominal Coagulation Parameter (Blood and lymphatic system disorders) | 1 (1)
Abdominal Lab Value (General disorders) | 2 (3)
Accelerated Idioventricular Rhythm (Cardiac disorders) | 1 (1)
Accelerated Junctional Rhythm (Cardiac disorders) | 1 (1)
Acrocyanosis (Cardiac disorders) | 1 (1)
Acute Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Otitis Media (Ear and labyrinth disorders) | 2 (2)
Acute Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic Drug Reaction (General disorders) | 1 (1)
Anesthesia Reaction (Injury, poisoning and procedural complications) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1)
Antidromic Reciprocating Tachycardia (Cardiac disorders) | 1 (1)
Antral Erosion (Gastrointestinal disorders) | 1 (1)
Aortic Root Dilation (Cardiac disorders) | 1 (1)
Aortic Valve Regurgitation and Insufficiency/Valvular Regurgitation Aortic Valve (Cardiac disorders) | 1 (1)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arterial Hypertension/Hypertension (Vascular disorders) | 5 (5)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Atelectasis (Injury, poisoning and procedural complications) | 15 (15)
Atrial Ectopic Beats and Rhythm / Premature Atrial Beats and Contractions (Cardiac disorders) | 22 (24)
Atrial Escape Beat (Cardiac disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 11 (12)
Atrial Flutter (Cardiac disorders) | 7 (7)
Atrial Tachycardia (Cardiac disorders) | 6 (6)
Aura (General disorders) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Bacteremia (Infections and infestations) | 1 (1)
Bacterial Infection of the Skin (Skin and subcutaneous tissue disorders) | 2 (2)
Behavioral Alterations (Psychiatric disorders) | 1 (1)
Biventricular Hypertrophy / Combined Ventricular Hypertrophy (Cardiac disorders) | 2 (2)
Bleeding (General disorders) | 19 (20)
Blurred Vision (Eye disorders) | 2 (2)
Borderline Prolongation of QT Interval (Cardiac disorders) | 1 (1)
Brachial Plexus Injury (Injury, poisoning and procedural complications) | 1 (1)
Broad QRS Complex Arrhythmias (Cardiac disorders) | 1 (1)
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Bruise/Purpura Simplex (Injury, poisoning and procedural complications) | 59 (62)
Cardiomegaly (Cardiac disorders) | 2 (3)
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 86 (96)
Chest Tightness (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 2 (3)
Chronic Renal Failure (Renal and urinary disorders) | 1 (1)
Common Cold / Upper Respiratory Tract Infection (Infections and infestations) | 8 (8)
Congestive Heart Failure (Cardiac disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Coronary Artery Anomaly (Vascular disorders) | 1 (1)
Coronary Artery Disease (Vascular disorders) | 2 (2)
Cough (General disorders) | 4 (4)
Decreased Appetite (General disorders) | 1 (1)
Decreased Exercise Tolerance (General disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
Dehydration (General disorders) | 2 (2)
Dental Trauma (General disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Device Embolization (Injury, poisoning and procedural complications) | 2 (2)
Diarrhea (General disorders) | 1 (1)
Diastolic Dysfunction (Cardiac disorders) | 1 (1)
Difficulty Catching Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dilated Main Pulmonary Artery (MPA) (Vascular disorders) | 1 (1)
Discomfort (General disorders) | 1 (1)
Diverticulitis (Gastrointestinal disorders) | 2 (2)
Dizziness (General disorders) | 17 (17)
Drug Rash (Skin and subcutaneous tissue disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (18)
EKG Abnormalities (Cardiac disorders) | 1 (2)
Echo Finding (Cardiac disorders) | 4 (4)
Edema (General disorders) | 5 (5)
Elective Surgery (Surgical and medical procedures) | 3 (3)
Emesis / Vomiting (Gastrointestinal disorders) | 25 (25)
Enlarged or Dilated Left Atrium (LA) (Cardiac disorders) | 1 (1)
Epididymitis (Reproductive system and breast disorders) | 1 (1)
Epistaxis (General disorders) | 18 (19)
Fainting / Blackout (General disorders) | 1 (1)
Fatigue / General Fatigue (General disorders) | 6 (6)
Febrile Seizures (General disorders) | 1 (1)
Fever (General disorders) | 11 (12)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
First Degree Heart / AV Block / Cardiac Arrhythmia / First Degree AV Block (Cardiac disorders) | 10 (10)
Foreign Bodies (General disorders) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3)
Gastrointestinal Illness (Gastrointestinal disorders) | 1 (1)
General Malaise (General disorders) | 1 (1)
Head and Neck Abscesses (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (General disorders) | 55 (56)
Heart Block (Cardiac disorders) | 3 (3)
Heart Failure (Cardiac disorders) | 1 (1)
Heart Murmur (Cardiac disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 2 (2)
Hematochezia (Gastrointestinal disorders) | 1 (1)
Hematoma (General disorders) | 27 (27)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Herpes Simplex (Infections and infestations) | 1 (1)
Hyperlipidemia (General disorders) | 1 (1)
Hypotension (Cardiac disorders) | 10 (10)
Hypothermia (General disorders) | 1 (1)
Incomplete Right Bundle Branch Block (Cardiac disorders) | 17 (17)
Increased Left Atrial Pressure (Cardiac disorders) | 2 (2)
Increased PR Interval (Cardiac disorders) | 1 (1)
Interventricular Conduction Delay (Cardiac disorders) | 1 (1)
Inverted T Wave (Cardiac disorders) | 1 (1)
Irregular Menstrual Period (General disorders) | 1 (1)
Irritability (General disorders) | 1 (1)
Junctional Escape Rhythm / Intermittent Junctional Rhythm (Cardiac disorders) | 6 (6)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Lacerations (General disorders) | 1 (1)
Left Axis Deviation (Cardiac disorders) | 3 (3)
Left Ventricular Hypertrophy (by EKG) (Cardiac disorders) | 1 (1)
Left Ventricular Hypertrophy (by Echo) (Cardiac disorders) | 4 (4)
Lightheadedness (General disorders) | 4 (4)
Long Q-T (Cardiac disorders) | 1 (1)
Low Back Pain (Cardiac disorders) | 1 (1)
Low/ Coronary Atrial Rhythm (Cardiac disorders) | 7 (7)
Lower Left Lobe Infiltrate (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Macular Degeneration (Eye disorders) | 1 (1)
Melena (Gastrointestinal disorders) | 2 (3)
Mid-Sternal Chest Pressure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Migraine (General disorders) | 27 (29)
Mitral Valve Prolapse (Cardiac disorders) | 2 (2)
Mitral Valve Regurgitation / Mitral Insufficiency (Cardiac disorders) | 7 (7)
Multiple Calcified Granulomata in the Lung Fields (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Nausea (General disorders) | 12 (12)
Nickel Allergy (General disorders) | 1 (1)
Non-Cardiac Chest Pain (General disorders) | 5 (6)
Non-Specific EKG Change (Cardiac disorders) | 2 (2)
Numbness (General disorders) | 6 (6)
Obstructive Sleep Apnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Orthostatic Hypertension (Cardiac disorders) | 4 (4)
Otitis Media (Ear and labyrinth disorders) | 2 (2)
Overhydration (General disorders) | 1 (1)
Pain (General disorders) | 14 (14)
Palpitations (Cardiac disorders) | 50 (53)
Panic Attack (Psychiatric disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Paroxysmal Atrial Fibrillation (Cardiac disorders) | 1 (1)
Paroxysmal Atrial Tachycardia (Cardiac disorders) | 1 (1)
Paroxysmal Supraventricular Tachycardia (Cardiac disorders) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 27 (27)
Pericarditis (Cardiac disorders) | 2 (2)
Peripheral Vascular Disease (Vascular disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Premature Ventricular Contraction (Cardiac disorders) | 8 (8)
Presyncope (Cardiac disorders) | 1 (1)
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary Nodule (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Venous Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Regular Narrow QRS Tachycardia / Supraventricular Tachycardias (Cardiac disorders) | 1 (1)
Residual Interatrial Communication (Cardiac disorders) | 1 (1)
Residual Shunt (Cardiac disorders) | 1 (1)
Respiratory Illness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Right Atrial Enlargement (Cardiac disorders) | 3 (3)
Right Axis Deviation (Cardiac disorders) | 7 (7)
Right Bundle Branch Block / Complete Right Bundle Branch Block (Cardiac disorders) | 3 (3)
Right Ventricular Conduction Delay (Cardiac disorders) | 4 (4)
Right Ventricular Hypertrophy (Cardiac disorders) | 4 (4)
Rotator Cuff Tear (Musculoskeletal and connective tissue disorders) | 2 (2)
ST Segment Changes (Cardiac disorders) | 1 (1)
ST-T-Wave Abnormality (Cardiac disorders) | 3 (3)
Seizure / Convulsions Epilepsy (Nervous system disorders) | 2 (2)
Sinus Arrhythmias (Cardiac disorders) | 7 (7)
Sinus Bradycardia / Sinus Bradycardia (Cardiac Arrhythmia) (Cardiac disorders) | 23 (23)
Sinus Tachycardia (Cardiac disorders) | 15 (15)
Sinusitis (General disorders) | 2 (2)
Skin Lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Snoring (General disorders) | 1 (1)
Sore Throat (General disorders) | 4 (4)
Strep Throat (General disorders) | 2 (2)
Stroke (Vascular disorders) | 1 (1)
Swelling (General disorders) | 1 (1)
Syncope (Cardiac disorders) | 3 (3)
T-Wave Abnormalities (Cardiac disorders) | 1 (1)
T-Wave Inversion (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombus (Cardiac disorders) | 1 (1)
Tingling (Nervous system disorders) | 1 (1)
Transient Ischemic Attack (Vascular disorders) | 1 (1)
Tremor (Nervous system disorders) | 2 (2)
Tricuspid Regurgitation/Tricuspid Insufficiency/Valvular Regurgitation: Tricuspid Valve (Cardiac disorders) | 2 (2)
Unsustained/Nonsustained Ventricular Tachycardia/Cardiac Arrhythmia (Cardiac disorders) | 2 (2)
Ureteral Dysfunction (Renal and urinary disorders) | 1 (1)
Urinary Calculi (Renal and urinary disorders) | 1 (1)
VASC Bleeding (Vascular disorders) | 2 (2)
VASC Bruise (Vascular disorders) | 1 (1)
VASC Hematoma (Vascular disorders) | 5 (5)
VASC Pain (Vascular disorders) | 5 (5)
VASC Pseudoaneurysm (Vascular disorders) | 2 (2)
Vaso Vagal Response (Nervous system disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 5 (5)
Viral Syndrome (Infections and infestations) | 1 (1)
Other (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No